CLINICAL TRIAL: NCT00594945
Title: A Phase 2a, Open-label,Proof -Of-Concept Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Intranasal Clonazepam in Adult Subjects With Epileptic Seizures
Brief Title: Study of Intranasal Clonazepam in Adult Subjects With Epileptic Seizures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 07-001
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Results first posted 2014-07-01 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-05

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Clonazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intranasal Clonazepam 2 mg (Experimental)
  Interventions: Drug: Clonazepam
- Intranasal Clonazepam 3 mg (Experimental)
  Interventions: Drug: Clonazepam
- Intranasal Clonazepam both Dose Groups 2 mg & 3 mg (Experimental)
  Interventions: Drug: Clonazepam

INTERVENTIONS:
Drug: Clonazepam — 1 Dose

SUMMARY:
Evaluate the safety and efficacy of intranasal Clonazepam in subjects with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of refractory epilepsy
* No Nasal conditions that would preclude the use of intranasal product

Exclusion Criteria:

* Subject with a clinical significant unstable medical abnormality
* Subject currently or regularly taking Clonazepam

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-12; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Benson, PhD, Study Director — Jazz Pharmaceuticals
Locations (6):
- United States (5):
  - Clinical Trials. inc., Little Rock, Arkansas
  - Mid-Atlantic Epilepsy & Sleep Center, Bethesda, Maryland
  - Columbia Comprehensive Epilepsy Center, Neurological Institute, New York, New York
  - Ohio State University, Columbus, Ohio
  - Neurological Clinic of Texas, PA, Dallas, Texas
- Tampere University Hospital, Tampere, Finland

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Based on preliminary PK data, the study was terminated early prior to achieving planned enrollment numbers.
  Cohort 1 was dosed at 2mg. Cohort 2 was dosed at 3mg. Two subjects participated in both Cohorts.
Groups:
- Intranasal Clonazepam 2 mg: Treatment administered to subjects during Cohort 1
- Intranasal Clonazepam 3 mg: Treatment administered to subjects during Cohort 2
- Intranasal Clonazepam Both Dose Groups 2 mg & 3 mg: Subjects who were administered 2 mg during Cohort 1 and then 3 mg during Cohort 2
Period: Cohort 1 / Treatment Period 1
Arm/Group | Intranasal Clonazepam 2 mg | Intranasal Clonazepam 3 mg | Intranasal Clonazepam Both Dose Groups 2 mg & 3 mg
Started | 4 | 0 | 2
Completed | 4 | 0 | 2
Not Completed | 0 | 0 | 0
Period: Cohort 2 / Treatment Period 2
Arm/Group | Intranasal Clonazepam 2 mg | Intranasal Clonazepam 3 mg | Intranasal Clonazepam Both Dose Groups 2 mg & 3 mg
Started | 0 | 3 | 2
Completed | 0 | 3 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: There were 9 subjects total and 2 subjects were enrolled in both Cohorts.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intranasal Clonazepam 2 mg | Intranasal Clonazepam 3 mg | Intranasal Clonazepam Both Dose Groups 2 mg & 3 mg | Total
Number analyzed (Participants) | 4 | 3 | 2 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (8.74) | 29.7 (7.37) | 45.0 (1.41) | 33.4 (9.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 2
  Male | 2 | 3 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 3 | 2 | 9
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 1 | 4
  Finland | 2 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Spikes and Sharp Waves, Relative Change From Baseline to Treatment Day (%).
Description: Summary of video EEG number of spikes and sharp waves. Over a 24 hour period.
Time Frame: Change from baseline to treatment day
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Intranasal Clonazepam 2 mg | Intranasal Clonazepam 3 mg
Number analyzed (Participants) | 6 | 5
percentage of baseline | -7.4 (35.12) | -26.1 (33.94)

ADVERSE EVENTS:
Arm/Group | Intranasal Clonazepam 2 mg | Intranasal Clonazepam 3 mg
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 6/6 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intranasal Clonazepam 2 mg (N=6) | Intranasal Clonazepam 3 mg (N=5)
Lacrimation increased (Eye disorders) | 2 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Tongue Ulceration (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 2 | 2
Thirst (General disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Drooling (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Parosmia (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 1 | 0
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hypoaesthesia Facial (Skin and subcutaneous tissue disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 0
Pallor (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other